CLINICAL TRIAL: NCT00978510
Title: Health Personnel and the Control of Tuberculosis in a Hospital Environment
Brief Title: Study of Health Personnel and the Assistance to Patients With Tuberculosis in Hospital Environment
Status: Completed | Type: Observational
Sponsor: Sociedade Cearense de Infectologia (Other)
Responsible Party: Roberto da Justa Pires Neto, Universidade Federal do Ceará - UFC
Other Study IDs: TB HGWA 2
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Tuberculosis; Health Care Professionals; Hospital Environment
Keywords: Tuberculosis; Disease transmission; Exposure to biological agents; Health personnel
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate in hospital environment the knowledge of the health care professionals about fundamental concepts on tuberculosis and the accomplishment to respiratory isolation practices for patients with pulmonary tuberculosis hospitalized in a public hospital in Fortaleza, Ceará, Brazil.

DETAILED DESCRIPTION:
A cross-sectional study of health care professionals using a study instrument with questions to evaluate the knowledge of basic concepts about tuberculosis. A retrospective study reviewing medical records of patients with suspected tuberculosis hospitalized in the units of Adult and Pediatric Clinics and in the Critical Care Unit in a general hospital in Fortaleza-CE.

ELIGIBILITY:
Inclusion Criteria:

* Health care professionals working in a public hospital (HGWA) in the units of Adult and Pediatric Clinics and in the Critical Care Unit in a general hospital in Fortaleza-CE

Exclusion Criteria:

* Health care professionals working in HGWA but in units other than Adult and Pediatric Clinics and in the Critical Care Unit

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health care professionals from a public hospital in Brazil
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2004-01; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto J Pires Neto, Principal Investigator — Universidade Federal do Ceará - UFC
Locations (1):
- Hospital Geral Dr. Waldemar Alcântara, Fortaleza, Ceará, Brazil